CLINICAL TRIAL: NCT06087445
Title: A User-friendly, Non-invasive Neuro-orthosis That Restores Volitionally Controlled Grasp Functions for SCI Survivors With Tetraplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Battelle Memorial Institute (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lauren Wengerd, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CDMRP-SC210277P1
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spinal Cord Injury
Keywords: cervical spinal cord injury; chronic SCI; functional electrical stimulation; electromyography; functional rehabilitation; biomarker

STUDY DESIGN:
Intervention Model Description: Participants with chronic cervical spinal cord injury will complete a 12-week intervention protocol (3x/week) in an outpatient setting where they will practice functional activities using their hand/forearm while wearing the NeuroLife EMG-FES Sleeve System. We will assess functional outcomes using standardized clinical measures at 6 timepoints (double baseline, 4 weeks, 8 weeks, post-intervention, and 4 weeks post-intervention).
Masking Description: We will have an independent outcome rater conduct assessments who is not involved in the intervention, however, because this is a single-arm trial there is no way to truly 'mask' the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NeuroLife EMG-FES Sleeve System (Experimental): The NeuroLife EMG-FES System is a completely non-invasive system (surface electrodes only, no implantable components) worn on the forearm of participants and has up to 160 electrodes that can record electromyography (EMG), or muscle activity, and also electrically stimulate (FES) muscles. Using this combined, closed-loop technology participants will complete a 12-week protocol with a study therapist practicing functional activities using their hand/forearm while wearing the NeuroLife EMG-FES Sleeve System.
  Interventions: Device: NeuroLife EMG-FES Sleeve System

INTERVENTIONS:
Device: NeuroLife EMG-FES Sleeve System — Participants will complete a 12-week training protocol (3x/week, 1-2 hours/session) which includes an activity-based upper extremity training paradigm where participants will complete multiple repetitions attempting functional tasks in different categories (grip, grip with rotation, pinch, and pinch with rotation) while using the closed-loop EMG-FES system on one forearm/hand. Each category includes ~10 functional tasks (e.g., grip - open a jar; pinch with rotation - nuts and bolts) that progressively increase in difficulty. Each session will include massed practice of 3 functional tasks (20-minute blocks for each task) with rest breaks as needed to avoid fatigue. Sessions will include ~60 minutes of task practice, but they may last 1-2 hours to account for setup time and rest breaks.

SUMMARY:
The goal of this pilot clinical study is to investigate the NeuroLife EMG-FES Sleeve System, a closed-loop approach to functional electrical stimulation, in adults (n=12) with chronic (>12 months) tetraplegia due to spinal cord injury. Briefly, the NeuroLife EMG-FES System is a completely non-invasive system (surface electrodes only, no implantable components) worn on the forearm which has up to 160 electrodes that can record electromyography (EMG), or muscle activity, and also electrically stimulate (FES) muscles. The main questions this study aims to answer are: 1) What is the safety, feasibility, and early efficacy of the NeuroLife EMG-FES system on upper extremity outcomes in chronic SCI survivors with tetraplegia, and 2) Can EMG be used as a biomarker of recovery over time in chronic SCI participants undergoing rehabilitation? Participants will complete an intensive, task-oriented rehabilitation protocol using the NeuroLife EMG-FES System (3x/week x 12 weeks) in an outpatient setting. We will assess functional outcomes using standardized clinical measures of hand and arm function at six timepoints.

DETAILED DESCRIPTION:
In our prior work, members of our study team found that residual, sub-movement threshold EMG signals can be measured reliably from the forearm of chronically paralyzed individuals with spinal cord injury (SCI) using the NeuroLife EMG-FES System, and that EMG can be used to discriminate multiple attempted hand movements to drive continuous control of functional electrical stimulation (FES). Briefly, the NeuroLife EMG-FES System is a completely non-invasive system (surface electrodes only, no implantable components) worn on the forearm of participants and has up to 160 electrodes that can record electromyography (EMG), or muscle activity, and also electrically stimulate (FES) muscles. This allows users to attempt a movement and, even in the absence of physical movement, the system can detect what they are trying to do and electrically stimulate the muscles they are attempting to use. We hypothesize that this ability to control the system with participant's own muscle signals will assist in improving and restoring hand function of SCI survivors with tetraplegia. Furthermore, preliminary studies have suggested the potential for motor-intention driven FES to promote functional recovery after system use. With the dual-purpose use as a functional orthosis and as a rehabilitation tool for restoration of hand function, the NeuroLife EMG-FES System is poised to transform the state of care for those with hand impairment due to SCI.

The overarching goal of this proposal is to investigate the safety, feasibility, and early efficacy of the NeuroLife EMG-FES system on upper extremity outcomes in chronic SCI survivors with tetraplegia. A pilot clinical trial will allow us to test the following aims: Aim 1. Determine the early efficacy of using the NeuroLife EMG-FES System as a functional orthosis to complete functional activities after 12 weeks of task practice using the system. Aim 2. Determine the early efficacy of using the NeuroLife EMG-FES System as a rehabilitation tool to improve sensorimotor function after 12 weeks of task practice using the system. Aim 3. Develop and establish EMG-based biomarkers of neuroplasticity and recovery after chronic SCI.

We plan to conduct a pilot clinical trial investigating the NeuroLife EMG-FES Sleeve System in adults (n=12) with chronic (>12 months) tetraplegia due to spinal cord injury. Briefly, the NeuroLife EMG-FES System is a completely non-invasive system (surface electrodes only, no implantable components) worn on the forearm of participants and has up to 160 electrodes that can record electromyography (EMG), or muscle activity, and also electrically stimulate (FES) muscles. Using this combined, closed-loop technology participants will complete a 12-week protocol with a study therapist practicing functional activities using their hand/forearm while wearing the NeuroLife EMG-FES Sleeve System. We will assess functional outcomes using standardized clinical measures at 6 timepoints (double baseline, 4 weeks, 8 weeks, post-intervention, and 4 weeks post-intervention). At these timepoints we will also collect high-definition EMG data using the NeuroLife EMG-only system to investigate the ability to use EMG as a biomarker of recovery over time in chronic SCI participants undergoing rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. age 22 years or older
2. sustained a chronic (>12 months) cervical SCI (AIS A, B, C, or D) and is currently medically stable
3. unable to grasp and manipulate objects to allow independent performance of activities of daily living (e.g., Tetraplegia)
4. retain voluntary ability to enact unilateral shoulder and elbow movements either independently or with a mobile arm support
5. Willing and able to attend study sessions in Columbus, Ohio for 12 weeks, 3x/week and all assessment sessions (4 weeks prior to and 4 weeks following 12-week intervention protocol)
6. able to provide informed consent.

Exclusion Criteria:

1. medical contraindications to FES (e.g., pacemaker or other implanted devices, uncontrolled seizure disorder, cancer or open wounds on hands)
2. severe, uncontrolled autonomic dysreflexia
3. comorbid medical condition that, in the opinion of the PI, that may impact participant safety or study results
4. severe upper extremity spasticity or contractures that prevent FES-evoked wrist and finger movements
5. ventilator dependent
6. pregnant or plan to become pregnant (females only)
7. actively participating in upper extremity rehabilitation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Toronto Rehabilitation Institute Hand Function Test (TRI-HFT) (Object Manipulation Subtest) | baseline to 4-week post-intervention follow-up
  Evaluation of object manipulation while simulating 10 ADL tasks.
Aim 2: Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP), v2 | baseline to 4-week post-intervention follow-up
  Gold standard for measuring neurologic recovery and hand function across sensation, strength, prehension ability, and prehension performance.
Aim 3: Grasp and Release Test (GRT) | baseline to 4-week post-intervention follow-up
  Measurement of EMG derived biomarkers while attempting movements from the GRT.

SECONDARY OUTCOMES:
Aim 1: Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP), v2 (Prehension Performance Subtest) | baseline to 4-week post-intervention follow-up
  Measures ability to perform ADL-based tasks using different grasps.
Aim 2: Spinal Cord Independence Measure (SCIM)-III | baseline to 4-week post-intervention follow-up
  Patient-reported ADL participation across 3 domains: self-care, respiration and sphincter management, & mobility.

OTHER OUTCOMES:
Expedited International Standards for Neurological Classification of SCI (E-ISNCSCI) | baseline to 4-week post-intervention follow-up
  Expedited International Standards for Neurological Classification of SCI (E-ISNCSCI) to determine neurologic level of injury and ASIA score.
Tetraplegia Upper Limb Activities Questionnaire (TUAQ) | baseline to 4-week post-intervention follow-up
  A 10-item, 5-response patient-reported outcome measure assessing performance and satisfaction with UE activities for individuals with tetraplegia.
Demographics/History | baseline
  Self-report: Age, SCI history, caregiver support, etc.
Grasp and Release Test (full) | from 4 weeks after enrollment and end of 12 weeks +/- 2 weeks treatment
  Evaluates hand function, specifically the ability to grasp, move, and release various objects.
Action Research Arm test (ARAT) | from 4 weeks after enrollment and end of 12 weeks +/- 2 weeks treatment
  Assesses upper limb function with grasp, grip, pinch, and gross motor movements through a series of timed tasks involving everyday objects
Goniometry | from 4 weeks after enrollment and end of 12 weeks +/- 2 weeks treatment
  Measures joint range of motion (ROM) using a goniometer.
Dynamometry | from 4 weeks after enrollment and end of 12 weeks +/- 2 weeks treatment
  Measures grip strength, using a handheld device called a dynamometer.
Pinch Gauge | from 4 weeks after enrollment and end of 12 weeks +/- 2 weeks treatment
  Measures pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Wengerd, PhD, Principal Investigator — Ohio State University; David Friedenberg, PhD, Principal Investigator — Battelle Memorial Institute; Peyton Miller, OTD, Study Director — Ohio State University
Locations (2):
- United States (2):
  - Battelle Memorial Institute, Columbus, Ohio
  - Ohio State University Wexner Medical Center (Columbus Campus, Dodd Hall, Martha Morehouse Medical Pavillion), Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT06087445/ICF_001.pdf